CLINICAL TRIAL: NCT03564093
Title: Intranasal Dexmedetomidine Sedation and Analgesia During Pediatric Emergency Room Procedures: Randomized Double-blinded Clinical Trial
Brief Title: Intranasal Dexmedetomidine Sedation and Analgesia During Pediatric Emergency Room Procedures
Acronym: INDEXER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Outi Peltoniemi, Adjunct Professor of Pediatric Intensive Care, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INDEXER
Record Dates: First submitted 2018-03-13; First posted 2018-06-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Pain; Anesthesia
Keywords: pediatrics; sedation; emergency room sedation; intranasal sedation; dexmedetomidine; intranasal dexmedetomidine; children; pediatric; pediatric sedation
MeSH Terms: conditions — Pain | interventions — Administration, Intranasal; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Experimental): 1µg/kg intranasal dexmedetomidine
  Interventions: Drug: Intranasal Drug
- Placebo (Placebo Comparator): 0,01ml/kg intranasal 4,5% saline
  Interventions: Drug: Intranasal Drug

INTERVENTIONS:
Drug: Intranasal Drug — 1µg/kg of dexmedetomidine is given 30 minutes prior to intravenous cannulation or lumbar puncture
  Other Names: Dexmedetomidine
  Arms: Dexmedetomidine
Drug: Intranasal Drug — Intranasal 4,5% saline is given as a placebo 30 minutes prior to intravenous cannulation or lumbar puncture
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The study objective is to determine if intranasal dexmedetomidine is a safe and effective sedative drug during small painful procedures in the pediatric emergency room. Patients of the pediatric emergency room at Oulu university hospital with any medical condition requiring a small painful procedure like i.v. cannulation or lumbar puncture are asked to join the investigator's study if they would seem to benefit from a sedative drug during the procedure. Patients are randomly assigned to treatment group receiving intranasal dexmedetomidine 1µg/kg and to placebo group receiving 4,5% saline solution. The primary outcome is the success of the procedure. Cardiovascular and respiratory effects, the pain experienced by the patient, sedation scores and duration of crying are also monitored.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 1-12 years at the Oulu University Hospital emergency room who would benefit from sedative medication during small painful procedures like i.v. cannulation or lumbar puncture are asked to take part in our study

Exclusion Criteria:

* Allergy to dexmedetomidine or any supplementary elements of the Dexdor®-solution
* II or III degree AV-blockage without pacemaker
* Uncontrollable hypotension
* Stroke
* Critically ill patients who are admitted to the PICU
* Patients with clear cardiac or respiratory dysfunction
* Lowered level of consciousness
* Patients with increased risk of apnoeic events due to neurologic or metabolic conditions or extreme obesity
* A single patient can only take part in this study once.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2025-03-14 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Success of the procedure | After the first attempt of the procedure. The procedure is attempted 30 minutes after the study drug administration.
  The success of the first attempt of the procedure (venous cannulation or lumbar puncture) is evaluated at the end of the first attempt of the procedure. Succesfulness of venous cannulation is tested by the doctor on call by flushing the cannula with saline. If the cannula works without complications the cannulation is successfull. Lumbar puncture is successfull if all the samples needed from the liquor are collected.

SECONDARY OUTCOMES:
The duration of the procedure | The time from the start of the first attempt of the procedure to the success of the procedure. The procedure is attempted 30 after the study drug administration. Time from the first needle puncture to ending the procedure is recorded.
  The duration of the procedure
Parents assessment of the patients pain during the procedure | Parents return a questionnaire within 2 hours after the study drug has been administered.
  Parents assessment of the patients pain during the procedure on a visual analog scale. Parents fill in a questionnaire after the procedure is done. Questionnaire is returned to the research doctor during the follow up period.
Patient pain VAS | The numerical value of VAS is asked in the end of the follow up period of 2 hours.
  Patients assessment of the experienced pain with Visual Analog Scale is asked in the end of the follow up period. Visual Analog Scale is a numerical value for the pain experienced by the patient ranging from 0 to 10.
Patient pain FLACC | Every 5 minutes from 15 minutes prior the study drug to 2 hours after the administration of the drug.
  Assessment of pain levels of the patient with FLACC-scores. Assessment is done by the study doctor. FLACC is abbreviation of Faces Legs Activity Crying and Consolability scale. FLACC ranges from 0 to 10 as 0 being no pain at all and 10 being the most pain possible.
Patient sedation level | Every 5 minutes from 15 minutes prior the study drug to 2 hours after the administration of the drug.
  Assessment of sedation levels of the patient with Comfort-B-scores. Assessment is done by the study doctor.Comfort-B is a sedation scale ranging from 6 to 30. The lower the score the more sedated a patient is.
Duration of crying | Duration of crying during the time period from 25 minutes after the study drug administration for 30 minute time period in which the procedure is anticipated to be done.
  Duration of the patients crying during and after the procedure. The duration of crying associated with the procedure is recorded in seconds and minutes.
Effectivity of the drug | The follow up period lasts 2 hours from the study drug administration.
  The parents are asked in the end of the follow up period whether they think the patient received the experimental drug or placebo
Blood pressure | Every 5 minutes from 15 minutes prior the study drug to 2 hours after the administration of the drug.
  The systolic, diastolic and mean blood pressures are measured by manometer in every 5 minutes.
Respiratory rate | Every 5 minutes from 15 minutes prior the study drug to 2 hours after the administration of the drug.
  Respiratory rate is assessed by capnometry continuously and the rate is documented in every 5 minutes.
Oxygen saturation | Every 5 minutes from 15 minutes prior the study drug to 2 hours after the administration of the drug.
  Oxygen saturation is measured by pulse oxymetry continuously and the rate is documented in every 5 minutes
Heart rate | Every 5 minutes from 15 minutes prior the study drug to 2 hours after the administration of the drug.
  Heart rate is measured by ECG continuously and the rate is documented in every 5 minutes
Attempts needed to complete the procedure | After the successful attempt of the procedure. The first attempt of the procedure is done 30 minutes after the study drug administration. The assessment is done within 2 hours of the administration of the study drug.
  The number attempts needed to complete the procedure is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Outi Peltoniemi, Principal Investigator — Oulu University Hospital
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No